CLINICAL TRIAL: NCT02971813
Title: Feasibility of a Social Media Intervention for Exercise Motivation and Cardiac Rehabilitation Adherence
Brief Title: A Social Media Intervention for Exercise Motivation and Cardiac Rehabilitation Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Sigma Theta Tau International Honor Society of Nursing (Other)
Responsible Party: Principal Investigator, Lee Anne Siegmund, Nurse Scientist, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-1456
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Diseases
Keywords: cardiac rehabilitation; social media; adherence; motivation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facebook group (Experimental): The Facebook group will receive peer support, education and provider support via social media.
  Interventions: Behavioral: Facebook
- Comparison group (Active Comparator): The comparison group will receive the same educational materials as the Facebook™ group but will receive it in handout form, or via email if the patient misses cardiac rehabilitation on a particular week.
  Interventions: Behavioral: Facebook

INTERVENTIONS:
Behavioral: Facebook — 1. Volunteers will be recruited during inpatient stay, or via phone call or in person after discharge and prior to beginning cardiac rehabilitation.
  2. Participants will be given a baseline BREQ-3 survey and a PNSE scale.
  3. Patients will be randomized to Facebook™ versus comparison groups using a blocked randomization.
  4. The Facebook™ intervention will include peer support, education, provider support and text message prompts when new posts are added.
     1. Educational posts will cover topics that will cover healthcare information.
     2. Provider support will be posted much like the educational posts.
  5. The data collection for this study will take place prior to beginning cardiac rehabilitation, at which time the participants will receive the BREQ-3 and PNSE surveys either in person or via email link.
  6. Post-testing will include a BREQ-3 and PNSE surveys and count of the number of sessions completed in a 3 month period of time.

SUMMARY:
While cardiac rehabilitation (CR) has been shown to be effective at improving cardiovascular disease (CVD), participation is generally poor. The current feasibility study, will evaluate the impact of a social media intervention on motivation for exercise and adherence to CR sessions. Participants will be randomly assigned to a Facebook™ group or an enhanced education comparison group. The intervention will include access to a private Facebook™ group in which participants will receive weekly educational posts, weekly provider support and have the opportunity to communicate with other cardiac rehabilitation patients. Patients in the comparison group will be given the same educational materials, but these will be supplied in email. Participants will be asked to fill out a pre-post motivational questionnaire and the total number of sessions attended at the end of 3 months will be tallied. This study is grounded in Self-Determination Theory (SDT) and utilizes the Behavioral Regulation in Exercise Questionnaire (BREQ-2), which is based on the SDT.

DETAILED DESCRIPTION:
There is no research that addresses the use of Facebook as a tool to affect autonomous motivation in cardiac rehabilitation.

The purpose of the current feasibility study is to determine the feasibility of using a Facebook intervention, providing education, peer support and provider support, to affect change in motivation and self-determination for exercise, and adherence to cardiac rehabilitation in patients with CHD during a 12-week Phase II cardiac rehabilitation program. It is hypothesized that:

1. Scores for motivation for exercise overall will increase for patients exposed to a Facebook intervention and across individual motivational subtypes (regulations) relative to a comparison group who receive educational handouts and emails.
2. Percentage of cardiac rehabilitation sessions attended will be higher relative to a comparison group who receive educational handouts and emails.
3. Engagement in the private Facebook group (number of "hits" and "likes") will predict number of cardiac rehabilitation sessions attended and the change in motivation. The feasibility of a larger trial will be based on sample size and participants' engagement in the Facebook group.

Methodology Design This is a prospective, randomized controlled pilot trial to evaluate the feasibility of using a social media intervention to affect change in motivation for exercise and adherence to cardiac rehabilitation.

Setting and Sample:

The setting for this study will be in the outpatient cardiac rehabilitation at the main campus of a large tertiary care center in Northeast Ohio and several satellite facilities in the region. All patients receive an individualized exercise prescription based on functional capacity at intake. Most patients will be able to attend up to 3 sessions per week for a total of 36 sessions.

All patients who are current and regular Facebook users, have qualified for cardiac rehabilitation (diagnosed with CHD), and are entering cardiac rehabilitation at the main campus or one of the regional satellite hospitals of this tertiary care center, will qualify to participate in the study prior to beginning Phase II cardiac rehabilitation. Current Facebook users were chosen . Regular use will be defined as logging onto Facebook at least 2 times in the last month. Inclusion criteria will include both men and women 18 years of age or older and live within 100 miles of the main campus of this tertiary care center. Participants must be able to read and understand English in order to complete the questionnaires: the Psychological Need Satisfaction in Exercise Scale (PNSE) [37] and the Behavioral Regulation in Exercise Questionnaire-3 (BREQ-3). There will be no exclusion based on secondary diagnosis; however, participants must be able to exercise well enough to qualify to take part in cardiac rehabilitation.

Measures:

Change in motivation for exercise, will be measured at baseline and post-intervention using the BREQ-3. The BREQ-3 is a 24 question validated instrument that measures forms of intrinsic and extrinsic regulation of exercise behavior and is based on self-determination theory. Psychometrics were completed for the BREQ-2 by Markland and Tobin. Cronbach's alpha reliabilities were: amotivation = 0.83, external regulation = 0.79, introjected regulation = 0.80, identified regulation = 0.73, and intrinsic regulation = 0.86. The BREQ-3 includes 5 additional questions in addition to those on the BREQ-2 and has a new subscale for integrated regulation [33]. The subscales (regulations) of the BREQ-3 are used to calculate a relative autonomy index (RAI). Each question is answered on a 5 point Likert scale (0-4) and represents one of the regulations. The regulations are weighted then summed to give a single score. The resulting index gives an indication of individual respondent's self-determination for exercise.

The RAI will place individual motivational subtypes or behavioral regulations on the self-determination continuum from amotivated (lacking intention to exercise) to intrinsically motivated (self-determined or autonomously motivated).

The PNSE will be used to assess need satisfaction with exercise. This scale was designed to assess the perception of psychological need satisfaction associated with self-determined motivation for exercise and consists of 18 items on a 6 point Likert scale, with 3 subscales measuring perceived competence, autonomy, and relatedness. The scale showed high internal consistency (Cronbach >0.90) [37].

The percentage of cardiac rehabilitation sessions attended will be measured at the time of cardiac rehabilitation completion or dropout. It will calculated by dividing the number of sessions attended in a 3 month period of time by the total number of sessions allowed by insurance, and multiplying by 100.

Facebook engagement, will be assessed by measuring the number of "likes" by individuals on the private Facebook group. "Likes" (the number of times a participant clicks "like" on any of the Facebook posts) will be counted and, along with "hits" will be used to examine the association between engagement in the intervention, and cardiac rehabilitation adherence and change in motivation. A post-intervention questionnaire will be given to determine number of "hits". The participants will be asked to circle the number of times they accessed the private Facebook group per week: 0, 1-5, 6-10, 11-15 or > 15 times. The questionnaire will also be used to collect qualitative data on participants' perceptions of the intervention, including whether they felt supported in their care, more in touch with providers, whether or not they chatted with other Facebook members and if the Facebook group affected their exercise behaviors. The questionnaire will use a Likert scale (1, "not at all"-5, "quite a bit") for all questions and a section for comments.

Patient characteristics will include key demographic variables (age, gender, race, employment, distance to cardiac rehabilitation, socioeconomic status), engagement (number of "hits" and "likes"), and key clinical variables (functional capacity as measured in METS,cardiac rehabilitation indication, hypertension, diabetes, hyperlipidemia and waist circumference), which will be obtained from the electronic medical record.

Data Collection Procedures:

Volunteers will be recruited from the main campus or regional satellite hospitals of this tertiary care center during their inpatient stay, at the intake visit for cardiac rehabilitation at the main campus and satellite facilities in the region, or via phone call after discharge and up to the first cardiac rehabilitation session. Volunteers will be screened for Facebook use and interest in the study, then an email link will be sent which will include an information sheet. The Facebook group will be private in the sense that those not in the group will not be able to see the content. Participants will be given a baseline BREQ-3 questionnaire and PNSE scale. Participants will then be randomized to Facebook versus comparison groups using blocked randomization.

Intervention. The Facebook intervention will include peer support, education, provider support. These interventions are designed to minimize pressure, offer choices, and allow for peer interaction, and positive feedback in order to provide support for competence, autonomy and relatedness. Competence will be supported with use of educational posts. Autonomy support will come from provider posts. Relatedness will be supported by peer interaction and engagement in the Facebook group.

Educational posts will cover topics that will encourage participants to practice preventive heart care. The educational portion of the intervention is designed to offer clear information and structure, thus supporting competence. The posts may be in the form of text, video and/or pictures and will include materials from the hospital's health library, the American Heart Association and the Center for Disease Control.

Provider posts will include topics such as motivational quotes, encouragement, reminders to exercise independently, and reminders to contact providers with questions. These postings are designed to promote a sense of choice and help participants feel that providers see them as having a unique frame of reference thus being autonomy-supportive. Providers will be nurses on the research team, exercise physiologists nurse practitioners and physicians. Provider support will also include links to provider health chats, in which patients can chat online with providers at set dates and times.

Peer interaction on Facebook will be as frequently as the participant chooses and will be monitored daily by the research team. Engagement in Facebook is designed to offer an opportunity for social inclusion and a sense of involvement.

The comparison group will receive the same educational and provider support materials as the Facebook group but will receive it via email. Both groups will have the opportunity for weekly education classes and typical peer interactions.

Upon cardiac rehabilitation completion or dropout, post-data will be collected. It is anticipated that this pilot will take up to one year and will be completed when 30 participants for each group have been obtained.

Data Analysis Statistical Methods. This is a feasibility study and the sample size obtained will determine if the study is appropriately powered to detect the desired effect size. Patient characteristics will be summarized group using frequencies and percentages for categorical factors, and means and standard deviations for continuous measures. In order to examine the primary outcome, differences in change in motivation between groups, overall motivation using the RAI from the BREQ-3 will be evaluated using analysis of covariance (ANCOVA) models. Mean differences with 95% confidence intervals for group differences will be presented. Multivariate analysis of variance models will be used to evaluate differences in the change across individual motivation subtypes (regulations), using the BREQ-3, between groups overall. If significant, separate ANCOVA models for each subtype will be fit. Similar models will be used to compare changes in needs satisfaction scores, overall and separately among the three subscales, between groups. Two-sample t-tests will be used to compare number of sessions completed. As a secondary analysis, the relationships between patient characteristics, "hits" and "likes", and the outcome variables RAI change, number of sessions, and needs satisfaction change will be examined using t-tests and Pearson correlations. The correlation between changes in RAI and needs satisfaction will also be evaluated. Analyses will be performed using SAS software (version 9.4; Cary, NC). An overall significance level of 0.05 will be assumed for all tests.

Sample Size. The investigators plan to enroll 30 patients in each group. In the first 9 months of 2016, cardiac rehabilitation at the main campus of this tertiary care center had approximately 170 patient intakes. It is assumed that there will be a similar number of patient intakes for a 9 month period in 2017. Based on Facebook participation rates for those over age 50 [21] and the high participation rates in previous research projects in this facility's cardiac rehabilitation, it is estimated that 40% may meet eligibility requirements and agree to participate. Allowing for use of the first 8 participants to establish the Facebook group, the estimated sample size would then be 60 total participants for randomization to study group who can then be included in analysis. With this sample size, there will be 86% power to detect large effect sizes (d=0.8) for our study outcomes [40]. The primary aim of this sample size determination is to evaluate whether the proposed intervention is feasible, and to estimate the differences that might exist so that a larger trial that would have adequate power to detect smaller differences could be designed based on what was learned in this pilot study. The sample size of 30 per group was chosen primarily to facilitate a large intervention group, since the value of the intervention is predicated upon interaction among the participants.

ELIGIBILITY:
Inclusion Criteria:

* All male and female patients who are current and regular Facebook™ users, 18 years of age or older, have qualified for cardiac rehabilitation (diagnosed with cardiovascular disease), and are entering cardiac rehabilitation at the Main Campus of the Cleveland Clinic, will qualify for the study.

Exclusion Criteria:

* Participants must be able to exercise to the extent that they can take part in cardiac rehabilitation, must live within 100 miles and must be able to read and speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Motivation | 12 weeks
  Measured using Behavioral Regulation in Exercise Questionnaire-3 (BREQ-3)
Needs Satisfaction | 12 weeks
  Psychological Needs Satisfaction in Exercise Scale (PNSE)

SECONDARY OUTCOMES:
Adherence | 12 weeks
  Number of cardiac rehabilitation sessions attended

CONTACTS AND LOCATIONS:
Overall Officials: Lee A Siegmund, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Facebook log in's and demographic variables as well as survey responses will be shared with the research team. This information will be shared using encrypted flash drives and computers and emails will be confidential. All responses from participants on the Facebook™ group will be assigned a number and all other identifying information will be removed for data analysis. Any data on paper will be kept in the PI's locked office in a locked filing cabinet. All electronic data will be stored on the PI's computer which requires password entry and in a folder accessible only to the PI and the research team.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 2/27/17 until after manuscript submission
Access Criteria: With permission of PI

REFERENCES:
- [Background] Coyan GN, Reeder KM, Vacek JL, Coyan GN, Reeder KM, Vacek JL. Diet and exercise interventions following coronary artery bypass graft surgery: a review and call to action. Phys Sportsmed. 2014 May;42(2):119-29. doi: 10.3810/psm.2014.05.2064. PMID 24875979
- [Background] Deci EL, Ryan RM. The support of autonomy and the control of behavior. J Pers Soc Psychol. 1987 Dec;53(6):1024-37. doi: 10.1037//0022-3514.53.6.1024. PMID 3320334
- [Background] Ryan RM, Deci EL. Intrinsic and Extrinsic Motivations: Classic Definitions and New Directions. Contemp Educ Psychol. 2000 Jan;25(1):54-67. doi: 10.1006/ceps.1999.1020. PMID 10620381
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Sanchis-Gomar F, Perez-Quilis C, Leischik R, Lucia A. Epidemiology of coronary heart disease and acute coronary syndrome. Ann Transl Med. 2016 Jul;4(13):256. doi: 10.21037/atm.2016.06.33. PMID 27500157
- [Background] Savage PD, Sanderson BK, Brown TM, Berra K, Ades PA. Clinical research in cardiac rehabilitation and secondary prevention: looking back and moving forward. J Cardiopulm Rehabil Prev. 2011 Nov-Dec;31(6):333-41. doi: 10.1097/HCR.0b013e31822f0f79. PMID 21946418
- [Background] Servey JT, Stephens M. Cardiac Rehabilitation: Improving Function and Reducing Risk. Am Fam Physician. 2016 Jul 1;94(1):37-43. PMID 27386722
- [Background] Thomas RJ, King M, Lui K, Oldridge N, Pina IL, Spertus J; ACCFAHA Task Force on Performance Measures. AACVPR/ACCF/AHA 2010 Update: Performance measures on cardiac rehabilitation for referral to cardiac rehabilitation/secondary prevention services: A report of the American Association of Cardiovascular and Pulmonary Rehabilitation and the American College of Cardiology Foundation/American Heart Association Task Force on Performance Measures (Writing Committee to Develop Clinical Performance Measures for Cardiac Rehabilitation). J Cardiopulm Rehabil Prev. 2010 Sep-Oct;30(5):279-88. doi: 10.1097/HCR.0b013e3181f5e36f. No abstract available. PMID 20808157
- [Background] Williams MA, Ades PA, Hamm LF, Keteyian SJ, LaFontaine TP, Roitman JL, Squires RW. Clinical evidence for a health benefit from cardiac rehabilitation: an update. Am Heart J. 2006 Nov;152(5):835-41. doi: 10.1016/j.ahj.2006.05.015. PMID 17070142
- [Background] Deci EL, Ryan RM. Intrinsic Motivation and Self-determination in Human Behavior. New York, NY: Plenum Press. 1985. ISBN: 978-1-4899-2273-1.
- [Background] deCharms R. Personal Causation. New York, NY: Academic Press. 1968. ISBN 13: 9780122085505.
- [Result] Balatsoukas P, Kennedy CM, Buchan I, Powell J, Ainsworth J. The Role of Social Network Technologies in Online Health Promotion: A Narrative Review of Theoretical and Empirical Factors Influencing Intervention Effectiveness. J Med Internet Res. 2015 Jun 11;17(6):e141. doi: 10.2196/jmir.3662. PMID 26068087
- [Result] Cadmus-Bertram L, Irwin M, Alfano C, Campbell K, Duggan C, Foster-Schubert K, Wang CY, McTiernan A. Predicting adherence of adults to a 12-month exercise intervention. J Phys Act Health. 2014 Sep;11(7):1304-12. doi: 10.1123/jpah.2012-0258. Epub 2013 Oct 31. PMID 24176780
- [Result] Cavallo DN, Tate DF, Ries AV, Brown JD, DeVellis RF, Ammerman AS. A social media-based physical activity intervention: a randomized controlled trial. Am J Prev Med. 2012 Nov;43(5):527-32. doi: 10.1016/j.amepre.2012.07.019. PMID 23079176
- [Result] Cavallo DN, Tate DF, Ward DS, DeVellis RF, Thayer LM, Ammerman AS. Social support for physical activity-role of Facebook with and without structured intervention. Transl Behav Med. 2014 Dec;4(4):346-54. doi: 10.1007/s13142-014-0269-9. PMID 25584083
- [Result] Cox NS, Alison JA, Button BM, Wilson JW, Holland AE. Feasibility and acceptability of an internet-based program to promote physical activity in adults with cystic fibrosis. Respir Care. 2015 Mar;60(3):422-9. doi: 10.4187/respcare.03165. Epub 2014 Nov 25. PMID 25425703
- [Result] Devi R, Powell J, Singh S. A web-based program improves physical activity outcomes in a primary care angina population: randomized controlled trial. J Med Internet Res. 2014 Sep 12;16(9):e186. doi: 10.2196/jmir.3340. PMID 25217464
- [Result] Ghashghaei FE, Sadeghi M, Marandi SM, Ghashghaei SE. Exercise-based cardiac rehabilitation improves hemodynamic responses after coronary artery bypass graft surgery. ARYA Atheroscler. 2012 Winter;7(4):151-6. PMID 23205048
- [Result] Irwin B, Kurz D, Chalin P, Thompson N. Testing the Efficacy of OurSpace, a Brief, Group Dynamics-Based Physical Activity Intervention: A Randomized Controlled Trial. J Med Internet Res. 2016 May 6;18(4):e87. doi: 10.2196/jmir.5342. PMID 27154301
- [Result] Joseph RP, Keller C, Adams MA, Ainsworth BE. Print versus a culturally-relevant Facebook and text message delivered intervention to promote physical activity in African American women: a randomized pilot trial. BMC Womens Health. 2015 Mar 27;15:30. doi: 10.1186/s12905-015-0186-1. PMID 25886945
- [Result] Karmali KN, Davies P, Taylor F, Beswick A, Martin N, Ebrahim S. Promoting patient uptake and adherence in cardiac rehabilitation. Cochrane Database Syst Rev. 2014 Jun 25;(6):CD007131. doi: 10.1002/14651858.CD007131.pub3. PMID 24963623
- [Result] Magnezi R, Bergman YS, Grosberg D. Online activity and participation in treatment affects the perceived efficacy of social health networks among patients with chronic illness. J Med Internet Res. 2014 Jan 10;16(1):e12. doi: 10.2196/jmir.2630. PMID 24413148
- [Result] Maher C, Ferguson M, Vandelanotte C, Plotnikoff R, De Bourdeaudhuij I, Thomas S, Nelson-Field K, Olds T. A Web-Based, Social Networking Physical Activity Intervention for Insufficiently Active Adults Delivered via Facebook App: Randomized Controlled Trial. J Med Internet Res. 2015 Jul 13;17(7):e174. doi: 10.2196/jmir.4086. PMID 26169067
- [Result] Martin BJ, Hauer T, Arena R, Austford LD, Galbraith PD, Lewin AM, Knudtson ML, Ghali WA, Stone JA, Aggarwal SG. Cardiac rehabilitation attendance and outcomes in coronary artery disease patients. Circulation. 2012 Aug 7;126(6):677-87. doi: 10.1161/CIRCULATIONAHA.111.066738. Epub 2012 Jul 9. PMID 22777176
- [Result] Napolitano MA, Hayes S, Bennett GG, Ives AK, Foster GD. Using Facebook and text messaging to deliver a weight loss program to college students. Obesity (Silver Spring). 2013 Jan;21(1):25-31. doi: 10.1002/oby.20232. PMID 23505165
- [Result] Ribeiro F, Oliveira NL, Silva G, Campos L, Miranda F, Teixeira M, Alves AJ, Oliveira J. Exercise-based cardiac rehabilitation increases daily physical activity of patients following myocardial infarction: subanalysis of two randomised controlled trials. Physiotherapy. 2017 Mar;103(1):59-65. doi: 10.1016/j.physio.2015.12.002. Epub 2015 Dec 25. PMID 27012822
- [Result] Struik LL, Baskerville NB. The role of Facebook in Crush the Crave, a mobile- and social media-based smoking cessation intervention: qualitative framework analysis of posts. J Med Internet Res. 2014 Jul 11;16(7):e170. doi: 10.2196/jmir.3189. PMID 25016998
- [Result] Valle CG, Tate DF, Mayer DK, Allicock M, Cai J. A randomized trial of a Facebook-based physical activity intervention for young adult cancer survivors. J Cancer Surviv. 2013 Sep;7(3):355-68. doi: 10.1007/s11764-013-0279-5. Epub 2013 Mar 27. PMID 23532799
- [Result] Zeng W, Stason WB, Fournier S, Razavi M, Ritter G, Strickler GK, Bhalotra SM, Shepard DS. Benefits and costs of intensive lifestyle modification programs for symptomatic coronary disease in Medicare beneficiaries. Am Heart J. 2013 May;165(5):785-92. doi: 10.1016/j.ahj.2013.01.018. Epub 2013 Mar 1. PMID 23622916
- [Result] Haakma I, Janssen M, Minnaert A. Understanding the Relationship Between Teacher Behavior and Motivation in Students with Acquired Deafblindness. Am Ann Deaf. 2016 Summer;161(3):314-26. doi: 10.1353/aad.2016.0024. PMID 27477039
- [Result] Siegmund LA, Naylor J, Bena J, McClelland M. The relationship between Metabolic Syndrome and adherence to cardiac rehabilitation. Physiol Behav. 2017 Feb 1;169:41-45. doi: 10.1016/j.physbeh.2016.11.005. Epub 2016 Nov 11. No abstract available. PMID 27840095
- [Result] Rawstorn JC, Gant N, Meads A, Warren I, Maddison R. Remotely Delivered Exercise-Based Cardiac Rehabilitation: Design and Content Development of a Novel mHealth Platform. JMIR Mhealth Uhealth. 2016 Jun 24;4(2):e57. doi: 10.2196/mhealth.5501. PMID 27342791
- [Result] Wilson PM, Rodgers WM, Loitz CC, Scime, G. "It's who I am…really!" The importance of integrated regulation in exercise contexts. Journal of Biobehavioral Research. 2006; 11(2), 79-104.
- [Result] Lindwall M, Ivarsson A, Weman-Josefsson K, Jonsson L, Ntoumanis N, Patrick H, Thogersen-Ntoumani C, Markland D, Teixeira P. Stirring the motivational soup: within-person latent profiles of motivation in exercise. Int J Behav Nutr Phys Act. 2017 Jan 14;14(1):4. doi: 10.1186/s12966-017-0464-4. PMID 28088208
- [Result] Thorup CB, Gronkjaer M, Spindler H, Andreasen JJ, Hansen J, Dinesen BI, Nielsen G, Sorensen EE. Pedometer use and self-determined motivation for walking in a cardiac telerehabilitation program: a qualitative study. BMC Sports Sci Med Rehabil. 2016 Aug 18;8:24. doi: 10.1186/s13102-016-0048-7. eCollection 2016. PMID 27547404
- [Result] Wilson P, Rogers WT, Rodgers WM. The Psychological Need Satisfaction in Exercise Scale. J Sport Exerc Psychol. 2006; 28, 231-51.
- [Result] Markland D, Tobin V. A modification of the Behavioral Regulation in Exercise Questionnaire to include an assessment of amotivation. Journal of Sport and Exercise Psychology. 2004; 26(2), 191-96. doi: 10.1123/jsep.26.2.191.
- [Result] Cocks K, Torgerson DJ. Sample size calculations for pilot randomized trials: a confidence interval approach. J Clin Epidemiol. 2013 Feb;66(2):197-201. doi: 10.1016/j.jclinepi.2012.09.002. Epub 2012 Nov 27. PMID 23195919
- [Derived] Siegmund LA, Bena JF, Morrison SL. Cardiac Rehabilitation Facebook Intervention: Feasibility Randomized Controlled Trial. JMIR Cardio. 2023 Jun 15;7:e46828. doi: 10.2196/46828. PMID 37318865
- [Derived] Siegmund LA, Ahmed HM, Crawford MT, Bena JF. Feasibility of a Facebook Intervention for Exercise Motivation and Cardiac Rehabilitation Adherence: Study Protocol. JMIR Res Protoc. 2017 Aug 18;6(8):e162. doi: 10.2196/resprot.7554. PMID 28821473
- See also: Pew Research — http://www.pewinternet.org/2015/10/08/social-networking-usage-2005-2015/
- See also: Exercise motivation measurement — http://pages.bangor.ac.uk/~pes004/exercise_motivation/scales.htm

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT02971813/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT02971813/ICF_001.pdf